CLINICAL TRIAL: NCT06657690
Title: The Efficacy and Safety of Irinotecan Liposome Combined with S-1 in PD-1/L1 Inhibitor Refractory Recurrent or Metastatic Nasopharyngeal Carcinoma: a Prospective, Single-arm Phase 2 Study
Brief Title: Irinotecan Liposome Combined with S-1 in PD-1/L1 Inhibitor Refractory Recurrent or Metastatic NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Professor, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.031
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma | interventions — irinotecan sucrosofate; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irinotecan liposome group (Experimental): Irinotecan liposome injection combined with S-1 every 4 weeks for up to 6 cycles, until intolerable toxicity, subject withdrawal of informed consent, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
  Interventions: Drug: Irinotecan liposome; Drug: S-1

INTERVENTIONS:
Drug: Irinotecan liposome — Irinotecan liposome injection, 50mg/m2, D1、D15, ivgtt, Q4w.
Drug: S-1 — S-1, D1-D14, BID, p.o., Q4w (BSA < 1.25 m2, 40 mg/dose; 1.25 m2 ⩽ BSA < 1.5 m2, 50 mg/dose; BSA ⩾ 1.5 m2, 60mg/dose).

SUMMARY:
This is a prospective, single-arm Phase 2 study to evaluate the efficacy and safety of Irinotecan Liposome injection combined with S-1 in patients with recurrent (unable to local curative treatment) or metastatic NPC who failed at least first-line anti-PD-1/L1.

DETAILED DESCRIPTION:
Fifty-six recurrent (unable to local curative treatment) or metastatic NPC patients who had failed at least first-line anti-PD-1/L1, whether or not combined with chemotherapy, were eligible to receive Irinotecan Liposome injection combined with S-1 for up to 6 cycles. All patients will be treated until disease progression as determined by the investigator based on RECIST 1.1 criteria, intolerable toxicity, subject withdrawal of informed consent, initiation of new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first. Regular visits and imaging examinations will be conducted to evaluate the efficacy and safety of the treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing to participate in the study, sign the informed consent form (ICF), and comply with study plan visits, treatment plans, laboratory tests, and other study procedures.

  2. Age ≥ 18 years. 3. Nasopharyngeal carcinoma confirmed by histopathology (differentiated or undifferentiated non-keratinous carcinoma).

  4. Recurrent or metastatic nasopharyngeal carcinoma that has failed at least first-line anti-PD-1/L1, whether or not combined with platinum-containing standard regimen (Anti PD-1/L1 exposure at least 6 weeks, and the protocol used at the time of enrollment in this study meets one of the following two points: (1) Relapse during adjuvant therapy after radiotherapy, or relapse within 6 months after the end of treatment; (2) First-line treatment phase, progression during anti-PD-1/L1 treatment, or progression within 3 months after the end of anti-PD-1/L1).

  5. Recurrent or metastatic nasopharyngeal carcinoma that is unable to local curative treatment (surgery or radiotherapy).

  6. At least one measurable lesion according to RECIST 1.1 criteria (the spiral CT scan diameter of the measurable lesion is ≥ 10 mm or the short diameter of the enlarged lymph node is ≥15mm ); lesions that have undergone local treatment can be selected as target lesions if there is clear evidence of significant progress compared to the end of treatment.

  7. ECOG PS (Eastern Cooperative Oncology Group Performance Status) score 0-1. Expected survival ≥3 months.

  8. Adequate main organ function: a. Liver function: AST and ALT ≤ 2.5 times ULN, bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert disease and serum bilirubin level ≤ 3 times ULN could be enrolled; patients with liver metastasis, ≤ 5 times ULN); b. Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 30 mL/min according to Cockcroft-Gault formula; c. Hematology: neutrophil absolute value (ANC) ≥1.0×10^9/L, hemoglobin (Hb) ≥ 9.0 g/dL, platelets ≥ 100×10^9/L.

Exclusion Criteria:

* 1. Severe allergy to Irinotecan liposome (such as systemic rash/erythema hypotension, bronchospasm, angioedema, or anaphylaxis).

  2.CYP3A4 strong inducer used within 2 weeks, or CYP3A4/UGT1A1 strong suppressor used within 1 week prior to initial administration.

  3. Estimated survival < 3 months. 4.HBsAg positive and HBV DNA copy number positive (quantitative detection ≥2000 IU/ml); Chronic hepatitis C blood screening positive (HCV antibody positive). Patients with normal liver function and concurrent antiviral therapy were determined by the investigator to be eligible for enrollment.

  5. HIV-positive people. 6. Patients with active bacterial infection, fungal infection, viral infection, or interstitial pneumonia require systemic treatment within 1 week prior to first administration.

  7. Received chemotherapy, targeted therapy, immunotherapy, or any investigational drug or other antitumor therapy within 4 weeks or 5 half-lives before first administration (whichever is shorter but at least 2 weeks).

  8. Received Chinese medicine with antitumor activity within 14 days before administration; Received other investigational drugs within 4 weeks prior to initial dosing.

  9. Patients who had undergone major surgery within 3 months prior to initial dosing or planned to undergo major surgery during the study period.

  10. Severe embolic events, such as cerebrovascular accidents (including transient ischemic attacks) and pulmonary embolism, occurred in the 6 months before screening.

  11. Diagnosed and/or treated with other malignancies within 2 years before initial administration (except for curable malignancies that have undergone radical treatment, such as skin basal cell, carcinoma in situ of the cervix, papillary thyroid cancer, etc).

  12. Severe cardiovascular disease during the 6 months before enrollment, including but not limited to the following: Acute myocardial infarction, unstable angina pectoris, coronary angioplasty or stenting, deep vein thrombosis, stroke; New York Heart Association Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%; According to the investigator's assessment, clinically significant abnormal electrocardiogram (ECG) at the time of screening.

  13. Pregnant or lactating women. 14. Serious dysfunction of heart, lung, liver, kidney, and other vital organs; serious and/or uncontrollable disease that may affect the patient's participation in the study (including, but not limited to, uncontrolled diabetes, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.).

  15. Other situations that the investigator determines to be inappropriate for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 1 year
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, an average of 1 year
  Progression-Free Survival PFS is defined as the duration from the date of treatment to progression or death
Overall survival (OS) | Through study completion, an average of 1 year
  Overall survival (OS) is defined as the duration from the date of treatment to death or last follow-up, with no restriction on the cause of death.
Incidence of adverse events | 1 year
  NCI-CTCAE 5.0 standard is adopted.

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth affiliated hosptial of Sun-yat Sen university, Zhuhai, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided